CLINICAL TRIAL: NCT04222764
Title: Evaluation of the Right Ventricular Systolic Function Using Real-time Three-dimensional Echocardiography in Intensive Care Unit Patients
Acronym: REA-3D-VD
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI19_0035 (REA-3D-VD)
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Ventricular Dysfunction, Right; Lung Diseases; Intensive Care Units
Keywords: Right ventricular failure; Lung Diseases; Intensive Care Units
MeSH Terms: conditions — Ventricular Dysfunction, Right; Lung Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Real-time three-dimensional echocardiography
  Interventions: Diagnostic Test: Real-time three-dimensional echocardiography

INTERVENTIONS:
Diagnostic Test: Real-time three-dimensional echocardiography — The initial hemodynamic assessment and monitoring using echocardiography will be performed within 12h following ICU admission. TTE will be performed systematically as first-line examination and TEE will be performed only on ventilated and sedated patients for whom additional information is required for their management, according to the standards of care of the participating centers. In that case, TEE will be performed immediately after TTE.
  3D echocardiographic measurements will be performed after the examination by two independent intensivists expert in critical care echocardiography who will be blinded from the usual parameters of RV systolic functions; these parameters will be measured during the examination to guide the management of patients, according to the standard of care of the participating centers.

SUMMARY:
Right ventricular failure (RVF) is an independent factor of mortality for many pulmonary diseases. Currently, RVF is defined as the incapacity of the RV to maintain the flow without dilating to use the Frank-Starling law (i.e., increase of the ejection volume associated to an increase of the preload). RVF is associated to RV systolic dysfunction which is conventionally defined as a decrease of the RV ejection fraction (RVEF) < 45%.

In the intensive care unit (ICU), acute RVF is mainly due to the acute respiratory distress syndrome (ARDS), sepsis or septic shock, and less often to severe pulmonary embolism or RV infarction.

The anatomical complexity of the RV precludes any geometrical assumption to estimate its volume, hence its ejection fraction (EF) using two-dimensional (2D) echocardiography. For this reason, the evaluation of RV systolic function is currently based on parameters used as surrogates of RVEF: fraction area change in 2D-mode, tricuspid annular plane systolic excursion (TAPSE) in M-mode, and maximal velocity of the systolic S' wave using tissue Doppler imaging.

Real-time three-dimensional (3D) echocardiography now enables accurate on-line measurement of RV volume and provides at the bedside the non-invasive assessment of RVEF. 3D transthoracic echocardiography (TTE) has been validated to measure RV volume and RVEF compared to MRI which is the gold standard. However, 3D transesophageal echocardiography (TEE) has not yet been validated in this specific clinical setting, while 2D TEE is frequently used in ICU in ventilated and sedated patients. Accordingly, the diagnostic ability of 3D echocardiography to quantify RV systolic function in ICU patients with RVF of any origin is currently unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old) hospitalized in the ICU and requiring echocardiography for any reason
2. With a disease at risk of being associated with RVF:

   * ARDS (Berlin definition)
   * Sepsis or septic shock (Sepsis-3 definition)
   * Pulmonary embolism
   * RV infarction
3. Affiliated to Social Security
4. Consent of the patient and/or his authorized representative to participate in the study.

Exclusion Criteria:

1. History of congenital cardiac disease
2. Patient under legal protection
3. Under any method of oxygen support or extracorporeal circulatory support (veno-venous extracorporeal membrane oxygenation, extracorporeal Life support...)
4. Non sinusal rhythm
5. Documented preexisting right cardiac disease
6. Quality of echocardiographic images incompatible with 3D assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: high risk right ventricular Failure intensive care patients
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Echocardiographic parameter | through study completion, an average of 28 days
  Agreement between the values of conventional echocardiographic parameters of RV systolic function and RVEF measured using TTE and considered as reference

SECONDARY OUTCOMES:
Threshold values of the conventional echocardiographic parameters identification | through study completion, an average of 28 days
  Threshold values of the conventional echocardiographic parameters to identify RV systolic dysfunction identified with RVEF measurement using 3D TTE (ROC curves: best sensitivity/specificity compromise)
RV end-diastolic volume measurement | through study completion, an average of 28 days
  RV end-diastolic measured using 3D TEE and 3D TTE (comparability if maximal difference < 10%)
RV end-systolic volume measurement | through study completion, an average of 28 days
  RV end-systolic volume measured using 3D TEE and 3D TTE (comparability if maximal difference < 10%)
RVEF measurement | through study completion, an average of 28 days
  RVEF measured using 3D TEE and 3D TTE (comparability if maximal difference < 10%)
RVEF measurement 3D | through study completion, an average of 28 days
  RVEF measured using 3D echocardiography (reference) and conventional echocardiographic parameters of RV systolic function in each disease responsible for RVF
Conventional echocardiographic parameters of RV systolic function measurement 3D | through study completion, an average of 28 days
  Conventional echocardiographic parameters of RV systolic function measured using 3D echocardiography in each disease responsible for RVF
Percentage of performed measurement | through study completion, an average of 28 days
  Percentage of performed measurements correlated to the theoretical number of possible measurements; intra and inter-observer reproducibility
Diagnosis of acute cor pulmonale | through study completion, an average of 28 days
  Agreement between conventional echocardiography and 3D echocardiography for the diagnosis of acute cor pulmonale (most severe type of RVF) as defined by an acute RV dilatation (RV/Left Ventricular end-diastolic area ratio > 0.6 in the long-axis view of the heart) associated to a paradoxical septum in the short-axis view of the heart
Number of deceased participant | through study completion, an average of 28 days
  ICU and hospital mortality
longitudinal systolic distortion of the RV free wall (strain) measurement | through study completion, an average of 28 days
  Relation and agreement between longitudinal systolic distortion of the RV free wall (strain), RVEF, and conventional parameters of RV systolic function

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Limoges university hospital, Limoges
  - CHU de TOURS, Tours